CLINICAL TRIAL: NCT07317011
Title: "Referral Attivo" Delta, Dallo Screening Alla Presa in Carico.
Acronym: HDV-Reflex
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: HDV Reflex
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis, Delta
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the "Active Delta Referral" Project is to estimate the prevalence of anti-HDV positivity among HBsAg-positive patients hospitalized in the Department of Medicine at ASST Papa Giovanni XXIII in Bergamo, as well as among patients at the SerD and the Prison Healthcare Unit of the same ASST, following the introduction of the new methodology in 2025, and to compare these findings with existing estimates for outpatients.

DETAILED DESCRIPTION:
Hepatitis Delta (HDV) is the most severe form of chronic viral hepatitis, associated with high morbidity and mortality, and affects only HBsAg-positive patients. Despite its severity, it remains largely underdiagnosed due to limited awareness among physicians and the absence of automatic screening. Current guidelines recommend testing all HBsAg-positive patients for anti-HDV, but in clinical practice this is rarely implemented.

The introduction of an "HDV-reflex" screening strategy, already successfully adopted in other countries, would allow for earlier identification of affected patients and improved clinical management, especially in light of the recent availability of new therapeutic options.

The HDV-reflex test will increase the number of patients screened for this virus, enabling an accurate estimate of HDV prevalence among HBV-positive individuals. It will also improve referral pathways and indications for antiviral treatment, and over time reduce the number of patients presenting at their first hepatology consultation with advanced HDV-related disease (such as HCC or decompensated liver disease requiring transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Hospitalized at the Department of Medicine of ASST Papa Giovanni XXIII in Bergamo, or attending the SerD or the Penitentiary Health Service of Bergamo.
* HBsAg positivity.
* Obtaining informed consent.

Exclusion Criteria:

* Lack of informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized (ward or day hospital) at the Department of Medicine of ASST Papa Giovanni XXIII in Bergamo (OMS square and San Giovanni Bianco facility), as well as outpatients attending the SerD and the Penitentiary Health Service of the same ASST, who are indicated for the HBsAg test, will undergo "active HDV referral." Patients who test positive for HBsAg between September 1, 2025, and August 31, 2026, and who provide informed consent, will be included in the study. For all patients, the Microbiology and Virology Laboratory will automatically perform the anti-HDV test and, in case of positivity, automatically perform the HDV RNA test, initiating referral to the Gastroenterology, Hepatology, and Transplantation Unit.
Sampling Method: Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of anti-HDV positive | At diagnosis during the baseline
  Estimate the percentage of anti-HDV positive individuals among HBsAg positive hospitalized patients

SECONDARY OUTCOMES:
HDV-positive patients | At diagnosis during the baseline
  Describe the main clinical characteristics of HDV-positive patients included in this study during 2025-2026.
HDV positivity data | At diagnosis during the baseline
  Compare the HDV positivity data from 2025-2026 with the data reported in the literature

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Sfreddo, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (3):
- Italy (3):
  - ASST PAPA GIOVANNI XXIII - Medicine Dept., Bergamo
  - ASST Papa Giovanni XXIII - SerD, Bergamo
  - ASST Papa Giovanni XXIII - SS Sanità Penitenziaria, Bergamo